CLINICAL TRIAL: NCT00957801
Title: Anabolic and Inflammatory Responses to Short-Term Testosterone Administration in Older Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-070
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2018-04-04 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Aging muscle; Androgen; Cytokines; Muscle metabolism
MeSH Terms: conditions — Sarcopenia | interventions — Testosterone; testosterone enanthate; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Testosterone injection (Active Comparator): Testosterone enanthate given as a single 100 mg Intramuscular (IM) injection
  Interventions: Drug: Testosterone injection
- Testosterone gel (Active Comparator): Testosterone topical gel (Androgel 1%) 10 mg administered daily for seven days
  Interventions: Drug: Testosterone gel
- Testosterone injection and Medrol 6 day dose pack (Active Comparator): Testosterone enanthate given as a single 100mg Intramuscular (IM) injection. Medrol 6 day dose pack was administered as directed with daily doses decreasing by 4mg per day with an additional 4mg given on day 7. Day one dose: 24mg, day two dose: 20mg, day three dose: 16mg, day four dose: 12mg, day five dose: 8mg, day six dose: 4 mg, day seven dose: 4mg.
  Interventions: Drug: Testosterone injection; Drug: Medrol
- Medrol 6 day dose pack (Active Comparator): Medrol 6 day dose pack was administered as directed with daily doses decreasing by 4mg per day with an additional 4mg given on day 7. Day one dose: 24mg, day two dose: 20mg, day three dose: 16mg, day four dose: 12mg, day five dose: 8mg, day six dose: 4 mg, day seven dose: 4mg.
  Interventions: Drug: Medrol

INTERVENTIONS:
Drug: Testosterone injection — 100 mg single IM injection
  Other Names: Testosterone enanthate
  Arms: Testosterone injection; Testosterone injection and Medrol 6 day dose pack
Drug: Testosterone gel — Testosterone gel 10 mg. administered topically daily for seven days
  Other Names: Androgel 1%
  Arms: Testosterone gel
Drug: Medrol — Medrol 6 day dose pack with an additional 4mg dose on day 7
  Other Names: methylprednisolone; Medrol dose pack
  Arms: Medrol 6 day dose pack; Testosterone injection and Medrol 6 day dose pack

SUMMARY:
Skeletal muscle loss is a common consequence of aging and in some individuals reaches a level that compromises health and quality of life. Age-associated increases in cytokine and inflammatory signaling may be important contributors to this process.

The investigators will assess the practical question of whether testosterone injection and gel application elicit similar responses. Resistance exercise will be used as a means of stimulating both inflammatory and anabolic responses in skeletal muscle. In order to assess the effects of testosterone on these responses, subjects will perform resistance exercise on two occasions separated by 7 days. The first session will be performed prior to the initiation of testosterone and/or medrol therapy and the second session will be performed after receiving therapy for 7 days.

DETAILED DESCRIPTION:
4 groups of healthy men aged 60 - 85 years were studied over 15 days, in 2 distinct time periods, pre-treatment and treatment.

Pre treatment week from study day -7 to study day -1. Treatment week from study day 1 to study day 8.

Groups:

1. Testosterone by injection (100mg testosterone enanthate) administered on study day 1.
2. Testosterone by gel application (10g/day Androgel 1%) administered daily beginning on study day 1 through study day 7.
3. Methylpredisone (Medrol) dose pack beginning on study day 1 (24mg) and decreasing by 4mg each day, with an additional 4mg taken on study day 7. Study day 1 (24mg), study day 2 (20mg), study day 3 (16mg), study day 4 (12mg), study day 5 (8mg), study day 6 (4mg), study day 7 (4mg).
4. Testosterone by injection (100mg testosterone enanthate) administered on study day 1 and Methylpredisone (Medrol) dose pack beginning on study day 1 (24mg) and decreasing by 4mg each day, with an additional 4mg taken on study day 7. Study day 1 (24mg), study day 2 (20mg), study day 3 (16mg), study day 4 (12mg), study day 5 (8mg), study day 6 (4mg), study day 7 (4mg).

Subjects were asked to fill out the Brief Fatigue Inventory daily for all 15 days.

Subjects were studied at the clinical research center before treatment (study day 1) and after treatment (study day 8). Resistance exercise was performed on study days 1 and 8. Blood was drawn before and after exercise for measurement of serum cortisol. Subjects were asked to return to the clinical research center each day during the treatment week (study days 1-8) for blood draws for measurement of total testosterone, estradiol and C-reactive protein (CRP). Labs were drawn on study days 1 and 8 for complete blood count, comprehensive metabolic panel and lipid panel.

Part 1:

In this part of the project we will study the acute response to testosterone treatment between two groups of subjects, comparing two methods of administration (injection vs. topical gel) in order to obtain pilot information for a subsequent, randomized, blinded long-term investigation.

Part 2:

In this part of the project we will study the acute response to Medrol (methylprednisolone) taken over 7 days with or without testosterone (given as 100mg IM) in order to obtain pilot information for a subsequent, randomized, blinded long-term investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60-85
* Gender: Male

Exclusion Criteria:

* Exclusionary medications will be an anticoagulant (Coumadin) because of the risk of bleeding during the biopsy procedure. Additional medications which will be disallowed for participation include: anabolic steroids, nitrates, antihistamines, and glucocorticoids.
* The subjects must be able to successfully complete an exercise stress test using the Bruce protocol . Subjects will be excluded without exercise testing, with a history of angina that occurs with exertion or at rest, or a myocardial infarction within the last 12 months. Subjects that demonstrate ³0.1 milliVolts (mV) horizontal or downsloping ST segment depression, a drop in systolic blood pressure of ³10 mm Hg, and/or frequent or repetitive arrhythmias (defined as ³10 premature ventricular contractions (PVC)/min, or couplets) during the stress test will be excluded.
* Subjects with LDL cholesterol above 200 mg/dL will be excluded .
* Any man with a history of breast cancer or prostate cancer, or any indication of an occult carcinoma from an elevation of prostate specific antigen (PSA) above 4.0 mg/L (53), or severe benign prostatic hypertrophy (BPH) by history (frequent urination, reduced stream) will be excluded.
* Subjects with liver dysfunction evidenced by a history of hepatitis B or hepatitis C, or by a three-fold elevation of liver enzymes (Alk phos, alanine aminotransferase (ALT), aspartate amino-transferase (AST) above normal on screening will be excluded from the study.
* Any subject with a blood pressure on three consecutive measurements taken at one week intervals that has a systolic pressure ³ 140 or a diastolic blood pressure ³ 90 will be excluded.
* Any subject who has a major medical illness such as diabetes, chronic obstructive pulmonary disease, or sleep apnea will be excluded. Moreover, subjects will not have a recent history of smoking tobacco. Morbidly obese older men (BMI > 35) will also be excluded.
* Subjects will evidence of kidney disease (serum creatinine > 2.0mg/dl) will be excluded from participation.
* Any subject with thyroid disease as determined by an abnormal thyroid stimulating hormone (TSH) level will be excluded from participation.
* Any subject testing positive for HIV will be excluded .
* Allergy to iodine, a component of Betadine which is used to prepare the subject's skin for invasive procedures, will be cause for exclusion from this study.
* Men with serum total testosterone concentrations greater than 500 ng/dL will be excluded.
* Subjects who engage in high intensity resistance training on a regular basis will be excluded.
* Subjects with a known coagulation disorder or with clinical evidence indicative of a bleeding disorder (easy bruising, "free bleeders") will not be enrolled in this study due to potential problems that could arise from muscle biopsy procedures.

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Urban, M.D., Principal Investigator — The University of Texas Medical Branch at Galveston
Locations (1):
- The University of Texas Medical Branch at Galveston, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 subjects screened, 15 subjects did not qualify, 2 subjects did not choose to participate. 29 subjects began the study and 28 subjects completed the study.
Groups:
- Testosterone Gel: Testosterone topical gel 10 mg administered daily for seven days
  Testosterone gel: Testosterone gel 10 mg. administered topically daily for seven days
Period: Overall Study
Arm/Group | Testosterone Injection | Testosterone Gel | Testosterone Injection and Medrol 6 Day Dose Pack | Medrol 6 Day Dose Pack
Started | 7 | 7 | 7 | 8
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Injection | Testosterone Gel | Testosterone Injection and Medrol 6 Day Dose Pack | Medrol 6 Day Dose Pack | Total
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (4) | 73 (5) | 73 (7.5) | 71 (7) | 72 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 7 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 7 | 6 | 7 | 8 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 7 | 7 | 6 | 7 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 7 | 8 | 29
Total Mass as Measured by DEXA [Mean (Standard Deviation); unit: kilograms] | 84.2 (82.83) | 89.6 (89.7) | 77.51 (76.93) | 89.04 (89.15) | 84.42 (15.8)
Lean Body Mass as measured by DEXA [Mean (Standard Deviation); unit: kilograms] | 52.60 (51.42) | 53.06 (52.66) | 49.22 (47.85) | 57.34 (57.84) | 52.77 (7.73)
Fat Mass as measured by DEXA [Mean (Standard Deviation); unit: kilograms] | 28.74 (28.64) | 33.32 (33.82) | 25.33 (26.12) | 28.40 (28.01) | 28.59 (9.99)

OUTCOME MEASURES:

1. Primary Outcome: Serum Total Testosterone Measured Before Treatment on Treatment Day 1 (Baseline Study)
Description: Testosterone was measured daily during the treatment week (treatment days 1 through 8). Serum testosterone was analyzed by UTMB clinical laboratory. Normal ranges are 72-623 ng/dL.
  Baseline testosterone was drawn before testosterone administration.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/dL | 307.57 (106.09) | 363.43 (95.76) | 408.17 (200.61) | 318.68 (129.68)

2. Primary Outcome: Serum Total Testosterone Measured on Treatment Day 2
Description: as for outcome 1
Time Frame: treatment day 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/dL | 980.86 (389.58) | 526.71 (127.59) | 191.87 (90.35) | 675.86 (316.83)

3. Primary Outcome: Serum Total Testosterone Measured on Treatment Day 3
Description: TTestosterone was measured daily during the treatment week (treatment days 1 through 8). Serum testosterone was analyzed by UTMB clinical laboratory. Normal ranges are 72-623 ng/dL.
  Baseline testosterone was drawn before testosterone administration.
Time Frame: treatment day 3
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/dL | 828.71 (375.94) | 527.43 (183.70) | 206.0 (89.35) | 673.29 (299.30)

4. Primary Outcome: Serum Total Testosterone Measured on Treatment Day 4
Description: as for outcome 1
Time Frame: treatment day 4
Population: One subject missed a testosterone monitoring visit for treatment day 4.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 6 | 7
ng/dL | 779.57 (399.73) | 441.71 (146.99) | 271.6 (134.93) | 734.57 (277.34)

5. Primary Outcome: Serum Total Testosterone Measured on Treatment Day 5
Description: TesTestosterone was measured daily during the treatment week (treatment days 1 through 8). Serum testosterone was analyzed by UTMB clinical laboratory. Normal ranges are 72-623 ng/dL.
  Baseline testosterone was drawn before testosterone administration.
Time Frame: treatment day 5
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/dL | 722.0 (302.10) | 460.14 (211.31) | 246.33 (131.30) | 669.71 (291.02)

6. Primary Outcome: Serum Total Testosterone Measured on Treatment Day 6
Description: as for outcome 1
Time Frame: treatment day 6
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/dL | 629.0 (272.56) | 536.43 (269.53) | 284.5 (166.0) | 645.14 (282.11)

7. Primary Outcome: Serum Total Testosterone Measured on Treatment Day 7
Description: as for outcome 1
Time Frame: treatment day 7
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/dL | 578.29 (173.58) | 485.86 (211.57) | 320.0 (113.06) | 579.57 (170.04)

8. Primary Outcome: Serum Total Testosterone Measured on Treatment Day 8 (Post Study)
Description: as for outcome 1
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/dL | 454.29 (57.12) | 435.14 (180.11) | 340.17 (127.27) | 481.14 (141.08)

9. Primary Outcome: Serum Estradiol Measured on Treatment Day 1 (Baseline Study)
Description: Estradiol was measured during the treatment week (treatment days 1 and 8). Serum estradiol was analyzed by UTMB clinical laboratory. Normal ranges are 20-47 pg/mL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
pg/mL | 22.86 (10.32) | 33.69 (17.04) | 36.33 (12.12) | 34.71 (10.95)

10. Primary Outcome: Serum Estradiol Measured on Treatment Day 8 (Post Study)
Description: as for outcome 9
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
pg/mL | 48.29 (12.20) | 33.43 (19.48) | 30.83 (7.05) | 47.14 (34.87)

11. Primary Outcome: Prostate Specific Antigen (PSA) Measured on Treatment Day 1 (Baseline Study)
Description: Prostate Specific Antigen (PSA) was measured before and after treatment week (study treatment days 1 and 8). PSA was analyzed by UTMB clinical laboratory. Normal ranges are less than 4.0 ng/mL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL | 1.92 (1.13) | 2.33 (1.60) | 1.85 (1.02) | 1.83 (1.25)

12. Primary Outcome: Prostate Specific Antigen (PSA) Measured on Treatment Day 8 (Post Study)
Description: as for outcome 11
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL | 1.98 (1.00) | 2.32 (1.64) | 1.78 (1.05) | 2.07 (1.60)

13. Primary Outcome: Hematocrit Measured on Treatment Day 1 (Baseline Study)
Description: Hematocrit was measured before and after treatment week (study treatment days 1 and 8). Hematocrit was analyzed by UTMB clinical laboratory. Normal ranges are 38.4% - 49.3%.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
percent | 39.17 (2.39) | 38.4 (3.71) | 40.45 (2.92) | 39.86 (2.33)

14. Primary Outcome: Hematocrit Measured on Treatment Day 8 (Post Study)
Description: as for outcome 13
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
percent | 38.74 (2.15) | 37.23 (3.57) | 40.53 (2.47) | 39.24 (2.72)

15. Primary Outcome: Total Cholesterol Measured on Treatment Day 1 (Baseline Study)
Description: Total Cholesterol was measured before and after treatment week (study treatment days 1 and 8). Total cholesterol was analyzed by UTMB clinical laboratory. Normal ranges are 120-200 mg/dL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 171.29 (35.72) | 165.57 (34.89) | 168.00 (24.51) | 156.71 (27.32)

16. Primary Outcome: Total Cholesterol Measured on Treatment Day 8 (Post Study)
Description: as for outcome 15
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 172 (46.45) | 162.86 (37.64) | 166.17 (23.57) | 141.86 (21.64)

17. Primary Outcome: Triglycerides Measured on Treatment Day 1 (Baseline Study)
Description: Triglycerides were measured before and after treatment week (study treatment days 1 and 8). Total cholesterol was analyzed by UTMB clinical laboratory. Normal ranges are 30-170 mg/dL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 140.42 (50.35) | 164.0 (44.45) | 122.5 (74.89) | 119.71 (35.04)

18. Primary Outcome: Triglycerides Measured on Treatment Day 8 (Post Study)
Description: as for outcome 17
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 112.57 (49.90) | 160.0 (58.91) | 155.17 (119.23) | 116.28 (22.94)

19. Primary Outcome: High-Density Lipoproteins (HDL) Measured on Treatment Day 1 (Baseline Study)
Description: High Density Lipoproteins (HDL) was measured before and after treatment week (study treatment days 1 and 8). HDL was analyzed by UTMB clinical laboratory. Normal ranges are higher than 35 mg/dL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 40.29 (6.29) | 38.86 (13.47) | 46.50 (8.94) | 42.14 (6.57)

20. Primary Outcome: High-Density Lipoproteins (HDL) Measured on Treatment Day 8 (Post Study)
Description: as for outcome 19
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 41.29 (9.60) | 36.71 (8.83) | 47.67 (5.35) | 43.43 (6.24)

21. Primary Outcome: Low-Density Lipoproteins (LDL) Measured on Treatment Day 1 (Baseline Study)
Description: Low Density Lipoproteins (LDL) was measured before and after treatment week (study treatment days 1 and 8). LDL was analyzed by UTMB clinical laboratory. Normal ranges are less than 160 mg/dL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 103.0 (27.76) | 93.57 (36.47) | 96.83 (18.24) | 90.71 (26.57)

22. Primary Outcome: Low-Density Lipoproteins (LDL) Measured on Treatment Day 8 (Post Study)
Description: as for outcome 21
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 104.0 (43.64) | 94.57 (40.61) | 87.5 (13.91) | 75.14 (19.79)

23. Primary Outcome: Very Low-Density Lipoproteins (VLDL) Measured on Treatment Day 1 (Baseline Study)
Description: Very Low Density Lipoproteins (VLDL) was measured before and after treatment week (study treatment days 1 and 8). VLDL was analyzed by UTMB clinical laboratory. Normal ranges are 5-60 mg/dL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 28 (10.13) | 33.14 (8.51) | 24.67 (14.99) | 23.86 (7.03)

24. Primary Outcome: Very Low-Density Lipoproteins (VLDL) Measured on Treatment Day 8 (Post Study)
Description: as for outcome 23
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 26.71 (8.50) | 29.29 (11.07) | 31.0 (24.02) | 24.71 (6.07)

25. Primary Outcome: C-Reactive Protein (CRP) Measured on Treatment Day 1 (Baseline Study)
Description: C-Reactive Protein (CRP) was measured during the treatment week (study treatment days 1 and 8). CRP was analyzed by UTMB clinical laboratory. Normal ranges are 0.0 - 0.8 mg/dL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 0.47 (0.23) | 0.33 (0.08) | 0.32 (0.4) | 0.4 (0.22)

26. Primary Outcome: C-Reactive Protein (CRP) Measured on Treatment Day 8 (Post Study)
Description: as for outcome 25
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
mg/dL | 0.47 (0.22) | 0.31 (0.04) | 0.32 (0.4) | 0.3 (0)

27. Primary Outcome: Dehydroepiandrosterone Sulfate (DHEA-S) Measured on Treatment Day 1 (Baseline Study)
Description: Dehydroepiandrosterone sulfate (DHEA-S) was measured before and after the treatment week on study treatment days 1 and 8. DHEA-S was analyzed by immunoassay on a Siemens Immulite 2000. Normal ranges are 28-290 ug/dL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ug/dL | 46.34 (48.14) | 34.16 (16.54) | 62.55 (53.20) | 46.07 (51.56)

28. Primary Outcome: Dehydroepiandrosterone Sulfate (DHEA-S) Measured on Treatment Day 8 (Post Study)
Description: as for outcome 27
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ug/dL | 37.96 (25.25) | 35.54 (14.52) | 34.74 (30.08) | 36.07 (35.77)

29. Primary Outcome: Sex Hormone Binding Globulin (SHBG) Measured on Treatment Day 1 (Baseline Study)
Description: Sex Hormone Binding Globulin (SHBG) was measured before and after the treatment week on study treatment days 1 and 8. SHBG was analyzed by immunoassay on a Siemens Immulite 2000. Normal ranges are 10-57 nmol/L.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
nmol/L | 21.78 (11.56) | 19.86 (8.51) | 25.66 (12.85) | 24.70 (9.63)

30. Primary Outcome: Sex Hormone Binding Globulin (SHBG) Measured on Treatment Day 8 (Post Study)
Description: as for outcome 29
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
nmol/L | 17.62 (4.8) | 20.13 (9.72) | 19.22 (11.71) | 14.57 (6.88)

31. Primary Outcome: Insulin Measured on Treatment Day 1 (Baseline Study)
Description: Insulin was measured before and after the treatment week on study treatment days 1 and 8. Insulin was analyzed by immunoassay on a Siemens Immulite 2000. Normal range is less than 25 uIu/mL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: uIu/mL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
uIu/mL | 8.53 (4.11) | 10.28 (8.09) | 4.09 (2.08) | 9.89 (10.0)

32. Primary Outcome: Insulin Measured on Treatment Day 8 (Post Study)
Description: as for outcome 31
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: uIu/mL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
uIu/mL | 7.47 (3.90) | 10.58 (7.13) | 3.92 (1.73) | 3.89 (1.80)

33. Primary Outcome: Insulin Like Growth Factor 1 (IGF-1) Measured on Treatment Day 1 (Baseline Study)
Description: Insulin like growth factor 1 (IGF-1) was measured before and after the treatment week on study treatment days 1 and 8. IGF-1 was analyzed by immunoassay on a Siemens Immulite 2000. Normal range is 33-220 ng/mL.
Time Frame: treatment day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL | 71.77 (33.99) | 69.2 (33.00) | 61.42 (40.36) | 90.74 (65.38)

34. Primary Outcome: Insulin Like Growth Factor 1 (IGF-1) Measured on Treatment Day 8 (Post Study)
Description: as for outcome 33
Time Frame: treatment day 8
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ng/mL | 80.16 (39.07) | 72.11 (26.20) | 69.17 (47.64) | 54.86 (47.34)

35. Primary Outcome: Cortisol Measured on Treatment Day 1 (Baseline Study) BEFORE Exercise Protocol
Description: Cortisol was measured before and immediately after the exercise protocol, before and after the treatment week on study treatment days 1 and 8. Serum Cortisol was analyzed by immunoassay on a Siemens Immulite 2000. Normal range is 5-25 ug/dL.
Time Frame: treatment day 1 - before exercise
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ug/dL | 7.25 (2.16) | 6.00 (1.67) | 6.64 (1.71) | 6.28 (1.61)

36. Primary Outcome: Cortisol Measured on Treatment Day 1 (Baseline Study) AFTER Exercise Protocol
Description: as for outcome 35
Time Frame: treatment day 1 - after exercise
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ug/dL | 7.71 (3.16) | 7.20 (2.71) | 4.76 (1.17) | 4.15 (1.64)

37. Primary Outcome: Cortisol Measured on Treatment Day 8 (Post Study) BEFORE Exercise Protocol
Description: as for outcome 35
Time Frame: treatment day 8 - before exercise
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ug/dL | 7.84 (3.13) | 5.97 (2.18) | 6.28 (2.90) | 5.19 (2.76)

38. Primary Outcome: Cortisol Measured on Treatment Day 8 (Post Study) AFTER Exercise Protocol
Description: as for outcome 35
Time Frame: treatment day 8 - after exercise
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
ug/dL | 7.05 (2.48) | 6.28 (3.41) | 4.40 (1.90) | 5.78 (2.38)

39. Primary Outcome: Global Fatigue Score as Measured by Brief Fatigue Inventory (BFI) in the Pre-treatment Week
Description: The Brief Fatigue Inventory is a 9 item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life), with "0" being no fatigue and "10" being as bad as you can imagine. The Global Fatigue score is calculated by averaging the answers of all the questions.
  This data is presented as the pre-treatment week average of study days -7 to -1.
Time Frame: Study days -7 to -1 (Pre - treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 7 | 7
units on a scale | 2.25 (0.41) | 1.47 (0.26) | 2.26 (0.37) | 1.86 (0.22)

40. Primary Outcome: Global Fatigue Score as Measured by Brief Fatigue Inventory (BFI) During the Treatment Week
Description: The Brief Fatigue Inventory is a 9 item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life), with "0" being no fatigue and "10" being as bad as you can imagine. The Global Fatigue score is calculated by averaging the answers of all the questions.
  This data is presented as the treatment week average of study days 1-8.
Time Frame: Study days 1-7 (treatment week)
Population: 1 subject did not complete the BFI during treatment week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone Injection | Testosterone Gel | Medrol 6 Day Dose Pack | Testosterone Injection and Medrol 6 Day Dose Pack
Number analyzed (Participants) | 7 | 7 | 6 | 7
units on a scale | 1.84 (0.30) | 1.79 (0.16) | 2.19 (0.48) | 1.57 (0.13)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Testosterone Injection | Testosterone Gel | Testosterone Injection and Medrol 6 Day Dose Pack | Medrol 6 Day Dose Pack
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No